CLINICAL TRIAL: NCT01840683
Title: An Open-label, Single Center Study to Evaluate the Efficacy and Safety of Heparin-induced Extracorporeal Lipoprotein Precipitation (H.E.L.P.) Therapy as a Treatment for Non-exudative (Dry) Age-related Macular Degeneration (AMD)
Brief Title: HELP Therapy for Dry AMD
Acronym: HELPuc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.Braun Avitum AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA-I-H-1202
Record Dates: First submitted 2013-04-05; First posted 2013-04-26 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Non-exudative (Dry) Age-related Macular Degeneration (AMD)
Keywords: Age-Related Macular Degeneration (AMD); Age Related Eye Disease Study (AREDS); Best-Corrected Visual Acuity (BCVA); Early Treatment Diabetic Retinopathy Study (ETDRS); Heparin-Induced Extracorporeal LDL-Cholesterol Precipitation (HELP); Visual Function Questionnaire (VFQ)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- H.E.L.P. therapy (H.E.L.P. Plasmat Futura System) (Experimental): A total of 8 apheresis therapies with the H.E.L.P. Plasmat Futura System will be performed over a period of 12 weeks.
  Interventions: Device: H.E.L.P. therapy (H.E.L.P. Plasmat Futura System)

INTERVENTIONS:
Device: H.E.L.P. therapy (H.E.L.P. Plasmat Futura System)
  Other Names: Heparin-Induced Extracorporeal LDL-Cholesterol Precipitation

SUMMARY:
This is an open-label, single center clinical investigation to evaluate the efficacy and safety of Heparin-induced Extracorporeal Lipoprotein Precipitation (H.E.L.P.) Therapy as a treatment for non-exudative (dry) Age-related Macular Degeneration (AMD). A total of 14 clinic visits are scheduled, one baseline visit, 8 visits for H.E.L.P. therapy treatments (to be performed over a period of 12 weeks for each patient) and 5 follow-up visits to be performed one week following the 4th H.E.L.P. therapy session and 12 weeks, 24 weeks, 36 weeks and 52 weeks after the final H.E.L.P. therapy session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-exudative (dry) AMD
* Male or female, between 50 and 90 years
* Presence of soft, confluent drusen in study eye
* At least one large (>125 μm) drusen
* Visual acuity (VA) between 20/32 and 20/100 Early treatment Diabetic Retinopathy Study (ETDRS) vision
* Fibrinogen level >100mg/dL
* Willing to continue lipid-lowering medication throughout the treatment phase if such medication was taken already before the study
* Willing to continue regular supplemental intake of Age related Eye Disease Study (AREDS) vitamins or comparable supplements throughout the study course
* Written informed consent

Exclusion Criteria (related to the underlying disease):

* Any evidence of wet AMD in either eye
* History of treatment for wet AMD in either eye
* Geographic atrophy involving fovea in study eye
* Fellow eye <20/400 VA
* Presence of cataract requiring treatment during study
* Presence of glaucoma requiring new treatment during study
* Presence of diabetic or other vascular retinopathy
* Previous retinal laser or surgical therapy
* Epiretinal membrane in study eye
* Any other ocular condition requiring therapy during the study

Exclusion Criteria (General):

* Participation in another clinical trial within 30 days
* Concurrent participation in another clinical trial
* Pregnancy or lactation
* Inability to give or understand informed consent
* Inability to maintain treatment and follow-up schedule
* Hypersensitivity to fluorescein
* Test positive for infectious status from HIV-, HBV- and HCV- infection

Exclusion Criteria (H.E.L.P. Apheresis):

* Heparin intolerance
* Heparin induced thrombocytopenia (HIT) II
* Hemorrhagic diathesis
* Ulcers in the gastrointestinal area
* Hemorrhage
* Coagulation disorder and neoplasm
* Liver diseases
* Severe heart failure and valvular defect
* Condition following apoplexia
* Dementia
* During pregnancy and lactation
* C1 esterase inhibitor deficiency or hereditary complement component 3 (C3) deficiency

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of H.E.L.P. therapy on the best corrected visual acuity (BCVA) in patients with non-exudative (dry) AMD. | Change from Baseline in the best corrected visual acuity (BCVA) at Week 24 after completion of H.E.L.P. therapy

SECONDARY OUTCOMES:
To evaluate the effects of H.E.L.P. therapy on the change in drusen area as assessed by colour photography. | Change from Baseline to Weeks 24 and 52 after completion of H.E.L.P. therapy
To evaluate the effects of H.E.L.P. therapy in area of abnormal autofluorescence as assessed by Fundus Autofluorescence (FAF). | Change from Baseline to Weeks 24 and 52 after completion of H.E.L.P. therapy
To evaluate the effects of H.E.L.P. therapy on overall visual functioning as assessed by the Visual Functioning Questionnaire (VFQ)-25 test. | Change from Baselineto Weeks 24 and 52 after completion of H.E.L.P. therapy
To evaluate the safety of H.E.L.P. therapy by assessing laboratory tests and vital signs. | Baseline and at all HELP therapy sessions being conducted after Baseline within 12 weeks.
To evaluate the effects of H.E.L.P. on the integrity of the outer retinal bands as assessed by Optical Coherence Tomography (OCT) | Change from Baseline in integrity of the outer retinal bands at Weeks 24 and 52 after completion of H.E.L.P. therapy
To evaluate the effects of H.E.L.P. therapy on the best corrected visual acuity (BCVA). | Change from Baseline to Week 52 after completion of H.E.L.P. therapy
To evaluate the effects of H.E.L.P. therapy on the AREDS severity scale as assessed by colour photography. | Change from Baseline to Weeks 24 and 52 after completion of H.E.L.P. therapy
To evaluate the effects of H.E.L.P. therapy on the incidence and change in area of geographic hypo autofluorescence as assessed by fundus autofluorescence images. | Change from Baseline to Weeks 24 and 52 after completion of H.E.L.P. therapy
To evaluate the effects of H.E.L.P. on the drusen volume as assessed by Optical Coherence Tomography (OCT) | Change from Baseline to Weeks 24 and 52 after completion of H.E.L.P. therapy
To evaluate the safety of H.E.L.P. therapy by assessing adverse events (AEs). | At all H.E.L.P. therapy sessions and follow-up visits being conducted after Baseline within 12 weeks and 12, 24, 36 and 52 weeks after completion of the H.E.L.P. therapy.
To evaluate the safety of H.E.L.P. therapy by physical examination. | At all H.E.L.P. therapy sessions being conducted after Baseline within 12 weeks and 52 weeks after completion of the H.E.L.P. therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Fareed Ali, MD, FRCS(C), Principal Investigator — Canadian Centre for Advanced Eye Therapeutics Inc.
Locations (1):
- Canadian Centre for Advanced Eye Therapeutics Inc., Mississauga, Ontario, Canada